CLINICAL TRIAL: NCT04638244
Title: Randomized Controlled Trial on Brief Online Music Intervention (BOMI) in Improving the Mental Well-being of Young People in the Community in Hong Kong
Brief Title: Brief Online Music Intervention (BOMI) in Improving the Mental Well-being of Young People in the Community in Hong Kong
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to work situation issue
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Chan Kai Tai, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KT0001
Record Dates: First submitted 2020-11-10; First posted 2020-11-20 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Mental Well-being
Keywords: Mental Well-being; Online Music; Young People; Randomized Controlled Trial
MeSH Terms: conditions — Psychological Well-Being | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOMI Group (Intervention Group) (Experimental): Listening to an expert-selected, theory-guided and self-chosen song each day actively in a personalized and focused way (Brief Online Music Intervention: BOMI) for 3 months
  Interventions: Behavioral: Music
- POM Group (Control Group) (Active Comparator): Receiving psychoeducational online message (POM) (for focused reading for 5 minutes) daily for 3 months
  Interventions: Behavioral: Reading messages

INTERVENTIONS:
Behavioral: Music — Brief Online Music
  Arms: BOMI Group (Intervention Group)
Behavioral: Reading messages — Reading psychoeducational messages
  Arms: POM Group (Control Group)

SUMMARY:
These unparalleled size, nature and complexity of youth mental health problems would leave a huge gap to fill after the Millennium, which would need stratified and timely interventions to improve the mental well-being and metal health of the youth in the general population. The use of music has been explored in improving the mental well-being and mental health in the young people. The progressively digitalized lifestyle of the youth as the digital natives is paralleled by frequent use of online music in their daily activities. This means that online music interventions can be a new, youth-friendly and accessible means to deliver interventions to the youth to improve their mental well-being and mental health. Therefore, it is worthwhile to further explore the potential as well as underlying mechanisms of online music in improving youth mental well-being and mental health in the community among young people as a population lifestyle strategy.

In this study, the investigators would conduct a Randomized Control Study on Brief Online Music Intervention (BOMI) by listening to a selected, guided and self-chosen online song each day actively in a personalized and focused way in improving the mental well-being of young people in the community. In the end, the possible design and promotion of specific, guided and evidence-based self-help brief online music intervention by listening to music daily as a lifestyle change can be an economic, convenient and evidenced-based mental well-being intervention strategy among the youth at a population level.

Aim: To study the effects of listening to an expert-selected, theory-guided and self-chosen online song each day actively in a personalized and focused way (Brief Online Music Intervention: BOMI) in improving mental well-being among young people in the community in Hong Kong Hypothesis: Listening to an expert-selected, theory-guided and self-chosen song each day actively in a personalized and focused way (Brief Online Music Intervention: BOMI) can improve mental well-being in the community among young people

DETAILED DESCRIPTION:
Introduction 75% of all mental disorders has onset before the age of 24, with pronounced effects extending throughout the lifespan. In recent years, studies showed that young people suffer from an overall poor mental well-being. A recent online community study in Hong Kong by the Department of Psychiatry of the University of Hong Kong shows that traumatic events, post-traumatic stress disorder and depressive symptom levels are significantly higher in young people under the age of 25.

These unparalleled size, nature and complexity of youth mental health problems would leave a huge gap to fill after the Millennium, which would need stratified and timely interventions to improve the mental well-being and mental health of young people in the general population.

As a fundamental component of youth culture in contemporary times, popular culture has intrinsic, spontaneous and interactive relationships with young people, who are at a developmental stage actively undergoing self-formation and socialization. Their relationships can vary widely, ranging from formation of styles and trends, self-regulation, emotion regulation, ideologies and attitudes, grouping and socializing, identification and even deep down to identity.

Among different forms of popular culture, music was said to be the most favoured leisure activity among adolescents. The use of music in engaging young people would be understandably considered to be direct, easy and effective, which should be a prerequisite for offering further help and interventions to improve the mental well-being and mental health of young people.

When it comes to the mental well-being and mental health of young people, the importance of music has been shown in prevention of mental health problems in young people as well as in facilitating those vulnerable young people receiving professional therapeutic supports. In addition, music has the potential to assist in achieving their optimal functioning and well-being.

To understand the pathway between culture and mind, progressive attempts have been made to explore the fundamental relationship between music, emotion and the brain. The evidence has been reviewed as a unified theory of musical emotions, ranging from 'everyday emotions' to 'aesthetic emotions', from a neuro-scientific approach.

To look back in the humankind history, music has been used for healing for millenniums, evolving in different forms and contents throughout generations. Last century, the emergence of popular music and popular songs was actually a reflection of the changing contemporary culture, economic conditions and ideologies. Across the millennium, the subsequent drastic digitalization in our world and daily living results in progressively digitalized lifestyle and habit of young people as the digital natives. In a recent global music report, 83% of people at the age of 16 to 24 have audio streaming engagement. This means that online music interventions can be a new, youth-friendly and accessible means to deliver interventions to young people to improve their mental well-being and mental health.

Therefore, it is worthwhile to further explore the potential as well as underlying mechanisms of online music in improving youth mental well-being and mental health in the community among young people as a population lifestyle strategy.

However, regarding to the exploration for such positive potential, despite that there is abundant evidence that young people can use music to improve mood daily, there is also evidence that inappropriate use of music for young people with psychological distress can cause negative effects on mental health. On the other hand, a study concluded that 'music is not causing problems, but rather reflecting and interacting with the young person's state of mental health'. In addition, it is more likely for young people to turn to media when they are in a negative mood. The lack of self-awareness may even play into music listening choices in young people in depression. Thus, it appears that there is a need to develop nuanced strategies for increasing awareness of the effect that music listening can have on young people's mood and well-being. In this regard, guidance based on theorizations and expert opinions would be a necessary part in designing any music interventions for young people in improving their mental well-being and mental health.

In terms of conceptualization and theorization, it is necessary to further delineate the possible factors and underlying mechanisms involved, through postulated interactions with rumination/reflection, resilience and self-esteem, in order to further provide evidence for specific music-based interventions in improving the well-being and mental health for young people.

In the end, the possible design and promotion of specific, guided and evidence-based self-help brief online music intervention by listening to music daily as a lifestyle change can be an economic, convenient and evidenced-based mental well-being intervention strategy among young people at a population level.

About ways of implementation, there is growing interest in studying automated music categorization for delivering the specific recommendations to music listeners, like by delineating a personalized music recommendation system based on electro-encephalography feedback. That means that people might be able to design recommendation algorithms with digital delivery tools in digital platforms based on evidence and guidance to deliver the desirable brief online music intervention conveniently in the population in future.

To go beyond, it is hoped that based on the findings, the investigators can further advocate evidence-based use of stratified online music interventions to improve the mental well-being and mental health in other aspects, like in clinical settings.

Methods The study is a randomized controlled trial (RCT) on Brief Online Music Intervention (BOMI) in improving the mental well-being of young people in the community by comparing participants receiving Brief Online Music Intervention (BOMI) daily for 3 months (BOMI Group) with participants receiving psychoeducational online message (POM) (for focused reading for 5 minutes) daily for 3 months (POM Group).

Study design The study is a parallel 3-months RCT of music-based intervention with 150 subjects to be randomized into the intervention group (BOMI Group) and 150 subjects to the control group (POM Group) as calculated below, with assessment at baseline and 3 months.

Sample Size Calculation The sample size was estimated using G*Power 3.1. Based on a previous meta-analysis on music-based intervention which reported a 0.545 effect size (16), the investigators anticipate our brief intervention will result in a smaller effect at 70% (i.e. 0.382). With 80% power and an alpha level of 5%, a sample size of 172 is required to detect the group difference. The target sample size is then inflated to 215 to allow for a 20% attrition rate, with 108 subjects on each arm. Based on this estimation, to increase the power further, the investigators have an estimation of 150 participants on each arm expected to be realistic to achieve in our study, with 20% loss to follow-up, leading to an available sample size of 120 on each arm and a total of 240 available subjects in the end.

Randomization Randomization would be carried out using a computer-generated sequence with a block size of 4 by an independent statistician. The statistician would advise the research assistant of allocations via encrypted e-mail; the research assistant then would notify participants by telephone.

Ethics Application to IRB would be made to the University of Hong Kong. Informed consent would be obtained and witnessed.

Protection against bias Participants are not blinded to the treatment allocation, as the intervention types are obvious. The research assistant enters data from the measures into computer. Once completed, an independent statistician would analyze the data; these would not be inspected until the end of the study.

Intervention

1. BOMI Group (Intervention Group) Development of the BOMI by an Expert Panel Firstly, the investigators would invite a group of psychiatrists, clinical psychologists, social workers, researchers, music therapists, music experts and musicians together with young people to form an expert panel to discuss about and formulate the guiding principles and therapeutic elements for subsequent respective song selections based on interdisciplinary consensus and conceptualisation frameworks.

   The guiding principles would be based on the identified four dimensions in linking music to well-being, namely relationship building, modifying emotions, modifying cognitions, emotional immersion.

   About the conceptualisation of the pathway of music in improving mental well-being, the postulated therapeutic elements would include engagement in structured and groovy music, ventilation with expressive music, distraction and relaxation with easy-listening music, sense of pleasurability with aesthetic music, narration in songs with sense of mastery and self worth through singing along, enhancement of interpersonal relationship with music sharing, as well as free improvisation with free association.

   About the postulated mechanisms of music in improving mental well-being, it would include changes in rumination/reflection, resilience and self-esteem.

   Their relationships with the expected outcome are tabulated in Figure 1 as attached.

   The expert panel members would also incorporate own individual taste, experience and expertise in selection of the songs, which would be even more appealing to young people.

   Based on these theorisations and postulations, the expert panel would choose songs to form a 'Me Mind Well' (MMW) Online Song Playlist on online streaming music platform specifically for young people in improving their mental well-being. The expert panel would also devise guiding tips for young people in choosing their own song appropriately by preventing possible negative effects and increasing their self-awareness, based on existing and further theorizations.

   Eventually, the Intervention Group (BOMI Group) subjects would choose a song each day according to the guidance, their mental state and preference to enter a five-minutes daily personalized and focused music space. Instruction would be given to the subjects to listen to their selected songs out of the MMW Online Song Playlist actively with full attention during the whole period.

   In view of the nature of the experience, there can be elements of mindfulness (i.e. awareness that arises through paying attention, on purpose, in the present moment, non-judgementally) in the intervention. In addition, a literature systemic review concluded that it seems that music listening can induce mindfulness states, with consequential benefits, e.g. improved attention or improved peak response intensity, which could also lead to improvement in mental well-being.
2. POM Group (Control group) Control Group (POM Group) subjects would receive psychoeducational online message (POM) (for focused reading for 5 minutes) daily for 3 months.

In essence, Intervention Group (BOMI Group) subjects would receive Brief Online Music Intervention (BOMI) daily for 3 months, while Control Group (POM Group) subjects would receive psychoeducational online message (POM) (for focused reading for 5 minutes) daily for 3 months.

Daily reminders would be sent by phone messages for the assigned tasks. They are requested to mark their finished tasks in calendar in digital form, which would be reviewed regularly by research assistants.

Assessment The assessments on music and pattern would be assessed at baseline and 3 months by a self-report questionnaire developed by the research team named Music Habit Questionnaire (MHQ).

The following assessments would be done at baseline and 3 months after completion of intervention by research assistants.

Primary outcome and measurement The primary outcome is mental well-being.

Measurement Tools:

Mental Well-Being: WHO 5

Secondary outcome and measurement Secondary outcomes include mental distress, mental health, musical engagement, mindfulness, QoL, rumination tendency, resilience and self-esteem

Measurement Tools:

Mental Distress: K6 Mental Health: Depression Anxiety Stress Scales (DASS) Musical Engagement: Healthy-Unhealthy Music Scale (HUMS) Mindfulness: Mindful Attention Awareness Scale QoL: 12-Item Short Form Survey (SF-12) (Mental Component score) Rumination: Rumination-Reflection Questionnaire (RRQ) Resilience: Connor-Davidson Resilience Scale (CD-RISC) Self-esteem: Rosenberg Self Esteem Scale (SES)

Qualitative Study Qualitative research in the Intervention Group (BOMI Group) about their experiences in engaging in a brief, regular, active, personalized and focused music space as a lifestyle habit by focus group interview with ethnographic approach would be conducted to analyze the subjective feelings and experiences, appreciation, cognitive appraisals, behavioural changes, emotional feelings, mindfulness, rumination, reflection, resilience, self-esteem, sociability and sense of mastery and pleasurability.

Data processing and analysis Primary Analysis The investigators would calculate Chi-square with 95% confidence intervals for dichotomous outcomes, and Paired t-test with 95% confidence intervals for changes in continuous outcomes. Repeat measure ANCOVA would also be used and appropriate statistical tests would be used for confounder adjustments. In particular, adjustment for mindfulness would also be performed to look into the possible confounding effect of mindfulness in mental well-being.

All tests would be two-tailed. After obtaining these results, the investigators would also calculate the standardised mean difference (Cohen's d) to facilitate interpretation of significance.

All analyses would be intention-to-treat. As a sensitivity analysis for the primary outcome, the investigators assume no change for those where the outcome is unobserved.

Secondary analysis The factors and underlying mechanisms involved, like postulated interactions between rumination, resilience and self-esteem along the pathway from music interventions to outcomes, are analyzed in the in the Intervention Group (BOMI Group) in order to further delineate evidence-based theories for the specific music-based interventions for young people. Multiple mediation analysis would be used.

ELIGIBILITY:
* Inclusion Criteria:

  1. No daily active, personalized and focused music listening in last 1 month (i.e. no daily self-chosen and personalized music listening with full attention)
  2. Living in community
* Exclusion criteria:

  1. Inability to access to internet and online music streaming platform daily
  2. No digital device with access to online music streaming platform

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Mental Well-being at 3 months | Baseline and 3 months
  WHO 5 (World Health Organization (Five) Well-being Index); score from 0 to 25; a higher score means a better result

SECONDARY OUTCOMES:
Change from Baseline Mental Distress at 3 months | Baseline and 3 months
  K 6 (Kessler Psychological Distress Scale); score from 0 to 24; a higher score means a worse result
Change from Baseline Mental Health at 3 months | Baseline and 3 months
  DASS (Depression Anxiety Stress Scales); score from 0 to 63; a higher score means a worse result
Change from Baseline Musical Engagement at 3 months | Baseline and 3 months
  HUMS (Healthy-Unhealthy Music Scale); HUMS healthy score from 5 to 25 with a higher score means a better result; HUMS Unhealthy score ranging from 8 to 40 with a higher score meaning a worse result
Change from Baseline Mindfulness at 3 months | Baseline and 3 months
  Mindful Attention Awareness Scale; score from 15 to 90; a higher score means a worse outcome
Change from Baseline Quality of Life at 3 months | Baseline and 3 months
  SF-12 (12-Item Short Form Survey) (Mental Component score); score 12 to 56; a higher score means a better outcome
Change from Baseline Rumination at 3 months | Baseline and 3 months
  RRQ (Rumination-Reflection Questionnaire); score from 24 to 120; a higher score means a worse outcome
Change from Baseline Resilience at 3 months | Baseline and 3 months
  CD-RISC (Connor-Davidson Resilience Scale); score form 0 to 40; a higher score means a better outcome
Change from Baseline Self-esteem at 3 months | Baseline and 3 months
  SES (Rosenberg Self-Esteem Scale); score from 4 to 40; a higher score means a worse outcome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Lonsdale AJ, North AC. Why do we listen to music? A uses and gratifications analysis. Br J Psychol. 2011 Feb;102(1):108-34. doi: 10.1348/000712610X506831. PMID 21241288
- [Background] Batt-Rawden KB, DeNora, T, Ruud E. Music listening and empowerment in health promotion: A study of the role and significance of music in everyday life of the long-term ill. Nordic Journal of Music Therapy 2005;14:20-136
- [Background] Gold C, Solli HP, Kruger V, Lie SA. Dose-response relationship in music therapy for people with serious mental disorders: systematic review and meta-analysis. Clin Psychol Rev. 2009 Apr;29(3):193-207. doi: 10.1016/j.cpr.2009.01.001. Epub 2009 Jan 22. PMID 19269725
- [Background] MacDonald R, Kreutz G, Mitchell L. What is music, health and wellbeing and why is it important? In R. MacDonald, G. Kreutz & L. Mitchell (Eds.), Music, Health, and Wellbeing. New York: Oxford University Press 2012;3-11.
- [Background] Juslin PN. From everyday emotions to aesthetic emotions: towards a unified theory of musical emotions. Phys Life Rev. 2013 Sep;10(3):235-66. doi: 10.1016/j.plrev.2013.05.008. Epub 2013 May 29. PMID 23769678
- [Background] Saarikallio S, Gold C, McFerran K. Development and validation of the Healthy-Unhealthy Music Scale. Child Adolesc Ment Health. 2015 Nov;20(4):210-217. doi: 10.1111/camh.12109. Epub 2015 May 18. PMID 26726295
- [Background] DeNora T. Music in Everyday Life. New York: Cambridge University Press. 2000
- [Background] McFerran K, Garrido S, O'Grady L, Grocke D, Sawyer SM. Examining the relationship between self-reported mood management and music preferences in Australian teenagers. Nord. J. Music Ther. 2015;24:1-17.
- [Background] Garrido S., Schubert E. Moody melodies: do they cheer us up? A study of the effect of sad music on mood. Psychol. Music. 2015;43:244-261.
- [Background] Garrido S., Schubert E. Music and people with tendencies to depression. Music Percept. 2015;32:313-321.
- [Background] Carpentier FR, Brown JD, Bertocci M, Silk JS, Forbes EE, Dahl RE. Sad Kids, Sad Media? Applying Mood Management Theory to Depressed Adolescents' Use of Media. Media Psychol. 2008 Jan 1;11(1):143-166. doi: 10.1080/15213260701834484. PMID 19768135
- [Background] Stewart J, Garrido S, Hense C, McFerran K. Music Use for Mood Regulation: Self-Awareness and Conscious Listening Choices in Young People With Tendencies to Depression. Front Psychol. 2019 May 24;10:1199. doi: 10.3389/fpsyg.2019.01199. eCollection 2019. PMID 31178806
- [Background] Chang HY, Huang SC, Wu JH. A personalized music recommnedation system based on electroencephalography feedback. Multimedia Tools and Application. 2017;76:19523-19542.
- [Background] de Witte M, Spruit A, van Hooren S, Moonen X, Stams GJ. Effects of music interventions on stress-related outcomes: a systematic review and two meta-analyses. Health Psychol Rev. 2020 Jun;14(2):294-324. doi: 10.1080/17437199.2019.1627897. Epub 2019 Jul 15. PMID 31167611
- [Background] Papinczak Z, Dingle GA, Stoyanov SR, Hides L. Young people's uses of music for wellbeing. Journal of Youth Studies. 2015 Feb;18(9).
- [Background] de la Cruz OL, Rodríguez-Carvajal R. Mindfulness and Music: A Promising Subject of an Unmapped Field. Int J Behav Res Psychol. 2014, 2(3), 27-35.
- See also: International Federation of the Phonographic Industry. Music Listening. 2019 — http://www.ifpi.org/wp-content/uploads/2020/07/Music-Listening-2019-1.pdf